CLINICAL TRIAL: NCT04973228
Title: A Phase 3, 8-Week, Parallel Group, Double Blind, Vehicle-Controlled Study of the Safety and Efficacy of ARQ-154 Foam 0.3% Administered QD in Subjects With Seborrheic Dermatitis
Brief Title: Trial of PDE4 Inhibition With Roflumilast (ARQ-154) Foam 0.3% for the Management of Seborrheic Dermatitis (STRATUM)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Arcutis Biotherapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ARQ-154-304
Record Dates: First submitted 2021-07-13; First posted 2021-07-22 (Actual); Results first posted 2024-03-12 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-02

CONDITIONS: Seborrheic Dermatitis
MeSH Terms: conditions — Dermatitis, Seborrheic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Roflumilast Foam 0.3% (Experimental): Participants with seborrheic dermatitis apply roflumilast foam 0.3% once daily (QD) for 8 weeks.
  Interventions: Drug: Roflumilast Foam
- Vehicle Foam (Placebo Comparator): Participants with seborrheic dermatitis apply vehicle foam QD for 8 weeks.
  Interventions: Drug: Vehicle Foam

INTERVENTIONS:
Drug: Roflumilast Foam — Roflumilast 0.3% foam for topical application
  Other Names: ARQ-154
  Arms: Roflumilast Foam 0.3%
Drug: Vehicle Foam — Vehicle foam for topical application
  Arms: Vehicle Foam

SUMMARY:
This phase 3, double-blind, vehicle-controlled study assessed the safety and efficacy of roflumilast (ARQ-154) foam 0.3% applied once daily (qd) for 8 weeks by participants with seborrheic dermatitis.

ELIGIBILITY:
Key Inclusion Criteria:

* Participants legally competent to sign and give informed consent and, if appropriate, assent as required by local laws.
* Males and females ages 9 years and older at the time of consent.
* Clinical diagnosis of seborrheic dermatitis of at least 3 months duration at Screening as determined by the Investigator. Stable disease for the past 4 weeks.
* Seborrheic dermatitis up to 20% BSA involvement. Involvement may be of the scalp and/or face and/or trunk and/or intertriginous areas.
* An Investigator Global Assessment (IGA) disease severity of at least Moderate ('3') at Baseline.
* Overall Assessment of Erythema and Overall Assessment of Scaling scores of at least Moderate ('2') at Baseline.
* Females of childbearing potential (FOCBP) must have a negative serum pregnancy test at Screening (Visit 1) and a negative urine pregnancy test at Baseline (Visit 2).
* Females of non-childbearing potential must either be post-menopausal with spontaneous amenorrhea for at least 12 months or have undergone surgical sterilization.
* Subjects in good health as judged by the Investigator.
* Subjects are considered reliable and capable of adhering to the Protocol and visit schedule according to the Investigator judgment.

Key Exclusion Criteria:

* Subjects who cannot discontinue treatment with therapies for the treatment of seborrheic dermatitis prior to the Baseline visit and during the study.
* Planned excessive exposure of treated area(s) to either natural or artificial sunlight, tanning bed or other LED.
* Previous treatment with ARQ-154 or ARQ-151.
* Subjects with any serious medical condition or clinically significant abnormality that would prevent study participation or place the subject at significant risk, as judged by the Investigator.
* Females who are pregnant, wishing to become pregnant during the study, or are breast-feeding.
* Subjects with a history of chronic alcohol or drug abuse within 6 months prior to Screening.
* Subjects, parent(s)/legal guardian(s) who are unable to communicate, read, or understand the local language(s).
* Subjects who are family members of the clinical study site, clinical study staff, or sponsor, or family members living in the same house of enrolled subjects.

Min Age: 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 457 (Actual)
Dates: Start 2021-07-08 (Actual); Primary Completion 2022-04-06 (Actual); Study Completion 2022-04-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Berk, MD, Study Director — Arcutis Biotherapeutics, Inc.
Locations (53):
- United States (43):
  - Arcutis Biotherapeutics Clinical Site 01, Scottsdale, Arizona
  - Arcutis Biotherapeutics Clinical Site 45, Encinitas, California
  - Arcutis Biotherapeutics Clinical Site 46, San Diego, California
  - Arcutis Biotherapeutics Clinical Site 64, San Diego, California
  - Arcutis Biotherapeutics Clinical Site 21, Santa Monica, California
  - Arcutis Biotherapeutics Clinical Site 42, Coral Gables, Florida
  - Arcutis Biotherapeutics Clinical Site 57, Delray Beach, Florida
  - Arcutis Biotherapeutics Clinical Site 33, Largo, Florida
  - Arcutis Biotherapeutics Clinical Site 31, North Miami Beach, Florida
  - Arcutis Biotherapeutics Clinical Site 65, Sanford, Florida
  - Arcutis Biotherapeutics Clinical Site 12, Tampa, Florida
  - Arcutis Biotherapeutics Clinical Site 10, Rolling Meadows, Illinois
  - Arcutis Biotherapeutics Clinical Site 03, Indianapolis, Indiana
  - Arcutis Biotherapeutics Clinical Site 22, Plainfield, Indiana
  - Arcutis Biotherapeutics Clinical Site 15, Louisville, Kentucky
  - Arcutis Biotherapeutics Clinical Site 04, Lake Charles, Louisiana
  - Arcutis Biotherapeutics Clinical Site 02, Rockville, Maryland
  - Arcutis Biotherapeutics Clinical Site 28, Rockville, Maryland
  - Arcutis Biotherapeutics Clinical Site 40, Clinton Township, Michigan
  - Arcutis Biotherapeutics Clinical Site 20, Detroit, Michigan
  - Arcutis Biotherapeutics Clinical Site 14, Fridley, Minnesota
  - Arcutis Biotherapeutics Clinical Site 44, Saint Joseph, Missouri
  - Arcutis Biotherapeutics Clinical Site 19, Reno, Nevada
  - Arcutis Biotherapeutics Clinical Site 34, East Windsor, New Jersey
  - Arcutis Biotherapeutics Clinical Site 66, New York, New York
  - Arcutis Biotherapeutics Clinical Site 63, The Bronx, New York
  - Arcutis Biotherapeutics Clinical Site 23, High Point, North Carolina
  - Arcutis Biotherapeutics Clinical Site 70, Winston-Salem, North Carolina
  - Arcutis Biotherapeutics Clinical Site 18, Bexley, Ohio
  - Arcutis Biotherapeutics Clinical Site 71, Portland, Oregon
  - Arcutis Biotherapeutics Clinical Site 08, Broomall, Pennsylvania
  - Arcutis Biotherapeutics Clinical Site 27, Pittsburgh, Pennsylvania
  - Arcutis Biotherapeutics Clinical Site 06, Knoxville, Tennessee
  - Arcutis Biotherapeutics Clinical Site 13, Arlington, Texas
  - Arcutis Biotherapeutics Clinical Site 11, Austin, Texas
  - Arcutis Biotherapeutics Clinical Site 41, College Station, Texas
  - Arcutis Biotherapeutics Clinical Site 60, Houston, Texas
  - Arcutis Biotherapeutics Clinical Site 26, Pflugerville, Texas
  - Arcutis Biotherapeutics Clinical Site 72, Plano, Texas
  - Arcutis Biotherapeutics Clinical Site 54, San Antonio, Texas
  - Arcutis Biotherapeutics Clinical Site 24, San Antonio, Texas
  - Arcutis Biotherapeutics Clinical Site 07, West Jordan, Utah
  - Arcutis Biotherapeutics Clinical Site 17, Norfolk, Virginia
- Canada (10):
  - Arcutis Biotherapeutics Clinical Site 35, Calgary, Alberta
  - Arcutis Biotherapeutics Clinical Site 37, Surrey, British Columbia
  - Arcutis Biotherapeutics Clinical Site 47, Winnipeg, Manitoba
  - Arcutis Biotherapeutics Clinical Site 43, Fredericton, New Brunswick
  - Arcutis Biotherapeutics Clinical Site 16, London, Ontario
  - Arcutis Biotherapeutics Clinical Site 29, Mississauga, Ontario
  - Arcutis Biotherapeutics Clinical Site 30, North Bay, Ontario
  - Arcutis Biotherapeutics Clinical Site 32, Peterborough, Ontario
  - Arcutis Biotherapeutics Clinical Site 36, Waterloo, Ontario
  - Arcutis Biotherapeutics Clinical Site 09, Westmount, Quebec

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were enrolled at 50 study centers in the US and Canada.
Groups:
- Roflumilast Foam 0.3%: Participants with seborrheic dermatitis applied roflumilast foam 0.3% once daily (QD) for 8 weeks.
- Vehicle Foam: Participants with seborrheic dermatitis applied vehicle foam QD for 8 weeks.
Period: Overall Study
Arm/Group | Roflumilast Foam 0.3% | Vehicle Foam
Started | 304 | 153
Completed | 276 | 138
Not Completed | 28 | 15
Not completed — Adverse Event | 2 | 3
Not completed — Lack of Efficacy | 1 | 3
Not completed — Lost to Follow-up | 12 | 4
Not completed — Withdrawal by Subject | 11 | 4
Not completed — Did not tolerate application | 1 | 0
Not completed — Wanted to early terminate and use own product | 0 | 1
Not completed — Missed visits due to new work schedule | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Roflumilast Foam 0.3% | Vehicle Foam | Total
Number analyzed (Participants) | 304 | 153 | 457
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.2 (16.81) | 41.8 (17.47) | 42.7 (17.03)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 151 | 78 | 229
  Male | 153 | 75 | 228
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 69 | 28 | 97
  Not Hispanic or Latino | 235 | 125 | 360
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4 | 0 | 4
  Asian | 18 | 10 | 28
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 36 | 15 | 51
  White | 234 | 122 | 356
  More than one race | 1 | 1 | 2
  Other | 11 | 4 | 15
Investigator Global Assessment (IGA) Baseline Score [Count of Participants; unit: Participants] — The IGA is 5-point scale assessing the severity of seborrheic dermatitis with total scores ranging from 0 ('clear') to 4 ('severe') [higher scores indicating greater severity].
  Participants
    2 - Mild | 0 | 0 | 0
    3 - Moderate | 287 | 141 | 428
    4 - Severe | 17 | 12 | 29
Worst Itch Numerical Rating Scale (WI-NRS) Baseline Score [Count of Participants; unit: Participants] — The WI-NRS is a simple, single-item scale to assess the participant-reported severity of this symptom, on a scale ranging from 0 ("no itch") to 10 ("worst imaginable itch") the participants experienced in the previous 24 hours (higher scores indicate higher itch severity). Population: Some participants did not have a baseline WI-NRS assessment.
  Participants
    0: number analyzed (Participants) | 297 | 152 | 449
    0 | 20 | 9 | 29
    1: number analyzed (Participants) | 297 | 152 | 449
    1 | 13 | 14 | 27
    2: number analyzed (Participants) | 297 | 152 | 449
    2 | 22 | 10 | 32
    3: number analyzed (Participants) | 297 | 152 | 449
    3 | 35 | 16 | 51
    4: number analyzed (Participants) | 297 | 152 | 449
    4 | 26 | 15 | 41
    5: number analyzed (Participants) | 297 | 152 | 449
    5 | 43 | 20 | 63
    6: number analyzed (Participants) | 297 | 152 | 449
    6 | 40 | 22 | 62
    7: number analyzed (Participants) | 297 | 152 | 449
    7 | 39 | 17 | 56
    8: number analyzed (Participants) | 297 | 152 | 449
    8 | 33 | 16 | 49
    9: number analyzed (Participants) | 297 | 152 | 449
    9 | 14 | 7 | 21
    10: number analyzed (Participants) | 297 | 152 | 449
    10 | 12 | 6 | 18

OUTCOME MEASURES:

1. Primary Outcome: Achievement of Success on the Investigator Global Assessment (IGA) at Week 8
Description: The percentage of participants achieving IGA "success" is presented. Success is defined as a score of 0 ('clear') or 1 ('almost clear') plus a 2-point improvement at Week 8. The IGA is 5-point scale assessing the severity of seborrheic dermatitis with total scores ranging from 0 ('clear') to 4 ('severe') [higher scores indicating greater severity].
Time Frame: Week 8
Population: All randomized participants are included.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Roflumilast Foam 0.3% | Vehicle Foam
Number analyzed (Participants) | 304 | 153
percentage of participants | 80 [74 to 84] | 58 [50 to 66]
Statistical Analysis 1: Comparison: Roflumilast Foam 0.3% vs Vehicle Foam; IGA Success at Week 8; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Stratified by pooled site and IGA strata with multiple imputation to handle missing data; Odds Ratio (OR) = 2.79, 95% CI 2-sided [1.75 to 4.45] — Stratified by pooled site and IGA strata with multiple imputation to handle missing data

2. Secondary Outcome: Achievement of Success in the Worst Itch Numeric Rating Scale (WI-NRS) at Week 8
Description: The percentage of participants achieving WI-NRS "success" is presented. The WI-NRS is a simple, single-item scale to assess the participant-reported severity of this symptom, on a scale ranging from 0 ("no itch") to 10 ("worst imaginable itch") the participants experienced in the previous 24 hours (higher scores indicate higher itch severity). The endpoint is the average of daily assessments reported during each study week, and requires at least 4 daily assessments reported during the week. In participants with a weekly average baseline pruritus score of ≥4, "success" is defined as achievement of a ≥4-point improvement from baseline in weekly average WI-NRS pruritus score at Week 8.
Time Frame: Week 8
Population: All randomized participants with a weekly baseline average WI-NRS score ≥4 are included.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Roflumilast Foam 0.3% | Vehicle Foam
Number analyzed (Participants) | 206 | 98
percentage of participants | 63 [56 to 70] | 41 [31 to 51]
Statistical Analysis 1: Comparison: Roflumilast Foam 0.3% vs Vehicle Foam; WI-NRS Success at Week 8; Test type: Superiority; p = 0.0001, Cochran-Mantel-Haenszel; Stratified by pooled site and IGA strata with multiple imputation to handle missing data; Odds Ratio (OR) = 2.95, 95% CI 2-sided [1.68 to 5.19] — Stratified by pooled site and IGA strata with multiple imputation to handle missing data

3. Secondary Outcome: Achievement of Success in the WI-NRS at Week 4
Description: The percentage of participants achieving WI-NRS "success" is presented. The WI-NRS is a simple, single-item scale to assess the participant-reported severity of this symptom, on a scale ranging from 0 ("no itch") to 10 ("worst imaginable itch") the participants experienced in the previous 24 hours (higher scores indicate higher itch severity). The endpoint is the average of daily assessments reported during each study week, and requires at least 4 daily assessments reported during the week. In participants with a weekly average baseline pruritus score of ≥4, "success" is defined as achievement of a ≥4-point improvement from baseline in weekly average WI-NRS pruritus score at Week 4.
Time Frame: Week 4
Population: All randomized participants with a weekly baseline average WI-NRS score ≥4 are included.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Roflumilast Foam 0.3% | Vehicle Foam
Number analyzed (Participants) | 206 | 98
percentage of participants | 48 [41 to 54] | 29 [21 to 39]
Statistical Analysis 1: Comparison: Roflumilast Foam 0.3% vs Vehicle Foam; WI-NRS Success at Week 4; Test type: Superiority; p = 0.0007, Cochran-Mantel-Haenszel; Stratified by pooled site and IGA strata with multiple imputation to handle missing data; Odds Ratio (OR) = 2.62, 95% CI 2-sided [1.47 to 4.67] — Stratified by pooled site and IGA strata with multiple imputation to handle missing data

4. Secondary Outcome: Achievement of Success in the WI-NRS at Week 2
Description: The percentage of participants achieving WI-NRS "success" is presented. In participants with a weekly average baseline pruritus score of ≥4, "success" is defined as achievement of a ≥4-point improvement from baseline in weekly average WI-NRS pruritus score at Week 2. The endpoint is the average of daily assessments reported during each study week, and requires at least 4 daily assessments reported during the week. The WI-NRS is a simple, single-item scale to assess the participant-reported severity of this symptom, on a scale ranging from 0 ("no itch") to 10 ("worst imaginable itch") the participants experienced in the previous 24 hours (higher scores indicate higher itch severity).
Time Frame: Week 2
Population: All randomized participants with a weekly baseline average WI-NRS score ≥4 are included.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Roflumilast Foam 0.3% | Vehicle Foam
Number analyzed (Participants) | 206 | 98
percentage of participants | 33 [27 to 40] | 16 [10 to 24]
Statistical Analysis 1: Comparison: Roflumilast Foam 0.3% vs Vehicle Foam; WI-NRS Success at Week 2; Test type: Superiority; p = 0.0016, Cochran-Mantel-Haenszel; Stratified by pooled site and IGA strata with multiple imputation to handle missing data; Odds Ratio (OR) = 2.74, 95% CI 2-sided [1.41 to 5.34] — Stratified by pooled site and IGA strata with multiple imputation to handle missing data

5. Secondary Outcome: Achievement of Success on the IGA at Week 2
Description: The percentage of participants achieving WI-NRS "success" is presented. The WI-NRS is a simple, single-item scale to assess the participant-reported severity of this symptom, on a scale ranging from 0 ("no itch") to 10 ("worst imaginable itch") the participants experienced in the previous 24 hours (higher scores indicate higher itch severity). The endpoint is the average of daily assessments reported during each study week, and requires at least 4 daily assessments reported during the week. In participants with a weekly average baseline pruritus score of ≥4, "success" is defined as achievement of a ≥4-point improvement from baseline in weekly average WI-NRS pruritus score at Week 2.
Time Frame: Week 2
Population: All randomized participants are included.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Roflumilast Foam 0.3% | Vehicle Foam
Number analyzed (Participants) | 304 | 153
percentage of participants | 43 [37 to 49] | 26 [19 to 33]
Statistical Analysis 1: Comparison: Roflumilast Foam 0.3% vs Vehicle Foam; IGA Success at Week 2; Test type: Superiority; p = 0.0002, Cochran-Mantel-Haenszel; Pooled by site and IGA strata with multiple imputation to handle missing data; Odds Ratio (OR) = 2.43, 95% CI 2-sided [1.54 to 3.84] — Pooled by site and IGA strata with multiple imputation to handle missing data

6. Secondary Outcome: Achievement of Success on the IGA at Week 4
Description: as for outcome 1
Time Frame: Week 4
Population: All randomized participants are included.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Roflumilast Foam 0.3% | Vehicle Foam
Number analyzed (Participants) | 304 | 153
percentage of participants | 73.1 [67.67 to 77.83] | 47.1 [39.19 to 55.10]
Statistical Analysis 1: Comparison: Roflumilast Foam 0.3% vs Vehicle Foam; IGA Success at Week 4; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Pooled by site and IGA strata with multiple imputation to handle missing data; Odds Ratio (OR) = 3.22, 95% CI 2-sided [2.06 to 5.03] — Pooled by site and IGA strata with multiple imputation to handle missing data

7. Secondary Outcome: Achievement of Overall Assessment of Scaling Score of 0 at Week 8
Description: The percentage of participants achieving Overall Assessment of Scaling score of 0 at Week 8 is presented. The Overall Assessment of Scaling is a simple, single-item scale to assess the subject-reported severity of this symptom, on a scale ranging from 0 ("No scaling: No scaling evident on lesions.") to 3 ("Severe: Coarse, thick scales, with flaking into clothes or skin."). Higher scores indicate greater symptom severity.
Time Frame: Week 8
Population: All randomized participants are included.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Roflumilast Foam 0.3% | Vehicle Foam
Number analyzed (Participants) | 304 | 153
percentage of participants | 58 [52 to 63] | 37 [29 to 45]
Statistical Analysis 1: Comparison: Roflumilast Foam 0.3% vs Vehicle Foam; Scaling Score of 0 at Week 8; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Stratified by pooled site and IGA strata with multiple imputation to handle missing data; Odds Ratio (OR) = 2.41, 95% CI 2-sided [1.56 to 3.73] — Stratified by pooled site and IGA strata with multiple imputation to handle missing data

8. Secondary Outcome: Achievement of Overall Assessment of Erythema Score of 0 at Week 8
Description: The percentage of participants achieving Overall Assessment of Erythema score of 0 at Week 8 is presented. The Erythema Assessment is a simple, single-item scale to assess the subject-reported severity of this symptom, on a scale ranging from 0 ("None: no evidence of erythema.") to 3 ("Severe: Intense [fiery red] erythema."). Higher scores indicate greater severity.
Time Frame: Week 8
Population: All randomized participants are included.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Roflumilast Foam 0.3% | Vehicle Foam
Number analyzed (Participants) | 304 | 153
percentage of participants | 58 [52 to 63] | 32 [25 to 40]
Statistical Analysis 1: Comparison: Roflumilast Foam 0.3% vs Vehicle Foam; Erythema Score of 0 at Week 8; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Stratified by pooled site and IGA strata with multiple imputation to handle missing data; Odds Ratio (OR) = 3.22, 95% CI 2-sided [2.05 to 5.06] — Stratified by pooled site and IGA strata with multiple imputation to handle missing data

ADVERSE EVENTS:
Time Frame: Up to ~8 weeks
Description: All randomized participants are included.
Arm/Group | Roflumilast Foam 0.3% | Vehicle Foam
All-Cause Mortality (participants affected / at risk) | 0/304 | 0/153
Serious Adverse Events (participants affected / at risk) | 1/304 | 0/153
Other Adverse Events (participants affected / at risk) | 0/304 | 0/153
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Roflumilast Foam 0.3% (N=304) | Vehicle Foam (N=153)
Keratoacanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor is supportive of publishing clinical trial findings. The process of coordinating publication efforts is detailed in the Clinical Trial Agreement.

DOCUMENTS (2):
  • Study Protocol (2022-05-05): https://cdn.clinicaltrials.gov/large-docs/28/NCT04973228/Prot_000.pdf
  • Statistical Analysis Plan (2022-09-22): https://cdn.clinicaltrials.gov/large-docs/28/NCT04973228/SAP_001.pdf